CLINICAL TRIAL: NCT04807517
Title: Buspirone for the Treatment of Anxiety in Williams Syndrome
Brief Title: Buspirone Treatment of Anxiety in Williams Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Robyn P. Thom, M.D., Assistant Professor of Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000376
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Williams Syndrome; Anxiety
MeSH Terms: conditions — Williams Syndrome; Anxiety Disorders | interventions — Buspirone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Buspirone (Experimental): Subjects will receive buspirone 2.5 mg each morning at the start of the trial. The dose will be increased by 2.5 mg per week in two divided doses daily depending on effectiveness and tolerability. The optimal dose will be reached by week 12 of treatment. The minimum starting dose will be 2.5 mg and the maximum total daily dose will be 30 mg. Medication will be dosed twice daily due to the short half-life (2-3 hours) of this medication.
  Interventions: Drug: Buspirone

INTERVENTIONS:
Drug: Buspirone — All participants in the study will receive open-label treatment with orally administered buspirone for the full duration of the 16-week trial. Buspirone has high affinity for serotonin 5-HT1A and 5-HT2 receptors and moderate affinity for dopamine D2 receptors. It is approved for the management of generalized anxiety disorder in adults.

SUMMARY:
The purpose of this study is to do a preliminary assessment of whether buspirone is effective, safe, and tolerable in the treatment of anxiety in children, adolescents, and adults with Williams syndrome.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients or their legal guardians giving written informed consent will be screened for study eligibility. Patients who meet the eligibility requirements will participate in a 16-week, flexibly-dosed, open-label trial of buspirone. The dose of buspirone will be adjusted over the first 12 weeks of the study and a stable dose will be maintained for the final four weeks of the trial. Adverse effects will be reviewed at each visit and standardized measures of anxiety will be conducted at weeks 4, 8, 12, and 16.

ELIGIBILITY:
Inclusion Criteria:

1. Age 5 to 65 years of age.
2. Diagnosis of WS confirmed via genetic testing or a clinical diagnosis made by a clinician with significant experience treating patients with WS.
3. Clinically significant anxiety as evidenced by a Pediatric Anxiety Rating Scale (PARS) score of 10 or greater (5-item scale). The PARS ("The Pediatric Anxiety Rating Scale (PARS): Development and psychometric properties." 2002) was chosen as an inclusion criterion (and outcome measure) since it assesses severity across common anxiety disorders in children including generalized anxiety, social anxiety, separation anxiety, and transition-associated anxiety. In addition, it is an instrument that allows the clinician to incorporate both child and parent report into a final clinician-rated score for each item.
4. A Clinical Global Impression Severity Item score ≥ 4 (moderate) for anxiety symptoms at Screen and Baseline.

Exclusion Criteria:

1. Diagnosis of OCD, posttraumatic stress disorder, major mood disorder, psychotic disorder, or substance use disorder. These disorders are exclusionary since the primary treatment of these disorders may require acute psychosocial treatments or other medications that would confound the assessments.
2. Presence of any past or present conditions that would make treatment with buspirone unsafe. This includes allergy to buspirone, liver or kidney disease, and pregnancy (or being sexually active without using acceptable methods to prevent pregnancy).
3. Use of selective serotonin reuptake inhibitors (SSRIs), serotonin norepinephrine reuptake inhibitors (SNRIs), benzodiazepines, antihistamines (as needed use of an antihistamine for the treatment of allergies will be permitted), or antipsychotics. Subjects will need to be off medications from these classes for at least 5 elimination half-lives prior to beginning the trial.
4. Use of other psychotropic medications which are ineffective, poorly tolerated, or sub-optimal in terms of dose. A board-certified child and adolescent psychiatrist will assess any other psychotropic medications being used and determine whether they are effective, tolerated, and optimal in terms of dose. Concurrent use of a psychotropic medication (other than SSRIs, SNRIs, benzodiazepines, antihistamines, or antipsychotics) will be allowed if the dose has been stable for 30 days and if they meet the criteria of effectiveness, tolerability, and dose.
5. Previous adequate trial of buspirone. An adequate trial will be defined as a total daily dose of ≥20 mg for at least 4 weeks. In addition, subjects who developed significant adverse effects during a trial of buspirone at any dose or duration will be excluded.
6. Severe or profound intellectual disability based on clinical assessment and review of standardized assessment of cognitive skills. Subjects will undergo standardized testing and be evaluated by study staff to determine cognitive capabilities. Participants determined to have severe or profound intellectual disability will be excluded.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robyn P Thom, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Lurie Center for Autism, Lexington, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between May 2021 and March 2023 through the Williams Syndrome Association and the Williams Syndrome Registry, as well as other specialty and primary care clinics. A recruitment letter was also sent to patients diagnosed with Williams Syndrome through the Mass General Brigham Patient Gateway secure online patient portal.
Pre-assignment Details: All 20 enrolled participants met inclusion criteria.
Period: Overall Study
Arm/Group | Buspirone
Started | 20
Started Taking Medication After Baseline | 19
Remained in Study at Week 12 | 18
Remained in Study at Week 16 | 18
Completed | 18
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Buspirone
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 17.4 [6 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean 16-Week Change in Pediatric Anxiety Rating Scale 5-Item Total Score
Description: The Pediatric Anxiety Rating Scale (PARS) is a clinician-rated instrument that assesses anxiety symptoms that are commonly associated with social anxiety, separation anxiety, and generalized anxiety disorders. Scaled score ranges from 0-25 with higher scores indicating more severe anxiety symptoms. Mean change was estimated using a repeated measures linear regression model with time in categories as the covariate and all non-missing scores for all measurement times as outcomes. A linear contrast estimated mean change between Baseline and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16; Change from Baseline to Week 16 reported
Population: All 20 participants contributed a baseline PARS 5-item total score to the analysis. Due to study discontinuation and a missing assessment, numbers of participants contributing post-baseline scores were 19 at week 4, 18 at week 8, 18 at week 12, and 18 at week 16.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Buspirone
Number analyzed (Participants) | 20
score on a scale | -7.9 [-10.0 to -5.9]
Statistical Analysis 1: Comparison: Buspirone; Test type: Other — Within-group test for 16-week change; p < 0.001, Regression, Linear; Repeated measures linear regression

2. Secondary Outcome: Proportion of Participants Who Responded to Treatment at 16 Weeks According to the Improvement Item of the Clinical Global Impression-Scale (Response Defined as CGI-I=1 or CGI-I=2)
Description: The Clinical Global Impressions Global Improvement (CGI-I) is designed to take into account all factors to arrive at an assessment of response to treatment. The CGI-I scale ranges from 1 to 7 (1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse), with lower scales indicating improvement (1=very much improved; 2=much improved). In this study, the CGI-I will be focused on the target symptom of anxiety. Participants with a CGI-I score of 1 or 2 will be classified as responders.
Time Frame: 16 weeks
Population: Participants who completed the study
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Buspirone
Number analyzed (Participants) | 18
Proportion of participants | 1.00 [0.82 to 1.00]

3. Secondary Outcome: Mean 16-Week Change in Child and Adolescent Symptom Inventory Anxiety-Modified Score
Description: The Child and Adolescent Symptom Inventory (CASI) is a caregiver completed questionnaire with items that map directly onto Diagnostic and Statistical Manual of Mental Disorders diagnostic criteria for anxiety disorders in children and adolescents. The CASI-Modified which includes 20 specific items that have been used to assess anxiety in subjects with developmental disabilities will be administered. Total score ranges from 0-20 with higher scores indicating more severe anxiety symptoms. Mean change was estimated using a repeated measures linear regression model with time in categories as the covariate and all non-missing scores for all measurement times as outcomes. A linear contrast estimated mean change between Baseline and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16; Change from Baseline to Week 16 reported
Population: All 20 participants contributed a baseline CASI modified score to the analysis . Due to study discontinuation and missing assessments, numbers of participants contributing post-baseline scores were 19 at week 4, 18 at week 8, 17 at week 12, and 18 at week 16.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Buspirone
Number analyzed (Participants) | 20
score on a scale | -8.9 [-12.8 to -4.9]

4. Secondary Outcome: Mean 16-Week Change in Screen for Childhood Anxiety Related Emotional Disorders Total Score
Description: The Screen for Childhood Anxiety Related Emotional Disorders (SCARED) includes both a child/self-report and parent-report form, each containing 41-items. It is used to screen for symptoms of panic disorder, separation anxiety disorder, social phobia, generalized anxiety disorder, and school phobia. Total score ranges from 0-82 and a total score of 25 or greater may indicate the presence of an anxiety disorder. Mean change was estimated using a repeated measures linear regression model with time in categories as the covariate and all non-missing scores for all measurement times as outcomes. A linear contrast estimated mean change between Baseline and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16; Change from Baseline to Week 16 reported
Population: All 20 participants contributed a baseline parent-report SCARED total score to the analysis . Due to study discontinuation and missing or incomplete assessments, numbers of participants contributing post-baseline parent-report scores were 19 at week 4, 18 at week 8, 17 at week 12, and 18 at week 16, and numbers contributing child-report scores were 9 at baseline, 8 at week 4, 10 at week 8, 7 at week 12, and 8 at week 16, with 10 contributing a score at either baseline or week 16.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Buspirone
Number analyzed (Participants) | 20
score on a scale
  Child/self-report form: number analyzed (Participants) | 10
  Child/self-report form | -16.0 [-28.1 to -3.9]
  Parent-report form | -9.3 [-13.4 to -5.1]

5. Secondary Outcome: Mean 16-Week Change in Each Subscale of the Aberrant Behavior Checklist
Description: The Aberrant Behavior Checklist (ABC-2) is a caregiver rated instrument that measures psychiatric symptoms and behavioral disturbance in subjects with developmental disability with 5 subscales. Each of its 58 items is scored on a 4-point scale (0=never a problem to 3=severe problem). The 5 subscales and their range of scores are: Irritability 0-45, with higher scores indicating more severe irritability; Social Withdrawal/Lethargy 0-48, with higher scores indicating more severe social withdrawal; Stereotypy 0-21, with higher scores indicating more severe stereotypy; Hyperactivity 0-48, with higher scores indicating more severe hyperactivity; Inappropriate Speech 0-12, with high scores indicating more severe inappropriate speech. Mean change was estimated using a repeated measures linear regression model with time in categories as the covariate and all non-missing scores for all measurement times as outcomes. A linear contrast estimated mean change between Baseline and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16; Change from Baseline to Week 16 reported
Population: All 20 participants contributed baseline ABC subscale scores to the analysis . Due to study discontinuation and missing assessments, numbers of participants contributing post-baseline scores were 19 at week 4, 18 at week 8, 17 at week 12, and 18 at week 16.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Buspirone
Number analyzed (Participants) | 20
score on a scale
  Irritability | -6.3 [-10.3 to -2.4]
  Social withdrawal/lethargy | -3.6 [-6.1 to -1.0]
  Stereotypy | -1.8 [-3.0 to -0.6]
  Hyperactivity | -6.2 [-9.4 to -2.9]
  Inappropriate speech | -0.8 [-1.7 to 0.1]

6. Secondary Outcome: Mean 16-Week Change in Pittsburgh Sleep Quality Index Global Score
Description: The Pittsburgh Sleep Quality Index (PSQI) questionnaire that will be completed by the subject's caregiver to assess sleep quality. The global score ranges from 0-21, where a higher score indicates greater sleep difficulty. Mean change was estimated using a repeated measures linear regression model with time in categories as the covariate and all non-missing scores for all measurement times as outcomes. A linear contrast estimated mean change between Baseline and Week 16.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16; Change from Baseline to Week 16 reported
Population: All 20 participants contributed a baseline PSQI global score to the analysis . Due to study discontinuation and missing assessments, numbers of participants contributing post-baseline scores were 19 at week 4, 18 at week 8, 16 at week 12, and 17 at week 16.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Buspirone
Number analyzed (Participants) | 20
score on a scale | -1.4 [-2.3 to -0.5]

ADVERSE EVENTS:
Time Frame: The earlier of 16 weeks or study discontinuation
Description: Adverse event data were collected via a structured side effect rating scale completed with the participant and their primary caregiver.
Arm/Group | Buspirone
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 19/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buspirone (N=20)
Diarrhea (Gastrointestinal disorders) | 8
Appetite decrease (General disorders) | 7
Stomach or abdominal discomfort (Gastrointestinal disorders) | 7
Nasal congestion or cold (Infections and infestations) | 6
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Sadness (Psychiatric disorders) | 5
Headache (Nervous system disorders) | 4
Flu or other respiratory problems (Infections and infestations) | 4
Dry mouth (General disorders) | 3
Interrupted sleep/ other sleep problems (Psychiatric disorders) | 3
Tiredness/fatigue (General disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Irritability (Psychiatric disorders) | 2
Sedation/drowsiness (General disorders) | 2
Weakness (General disorders) | 2
Dizziness/faintness (Nervous system disorders) | 1
Asthmatic symptoms (Respiratory, thoracic and mediastinal disorders) | 1
Appetite increase (General disorders) | 1
Indigestion (Gastrointestinal disorders) | 1
Localized rash (Skin and subcutaneous tissue disorders) | 1
Sweating (General disorders) | 1
Change in speech (Psychiatric disorders) | 1
Confusion (Nervous system disorders) | 1
Disinhibition (Psychiatric disorders) | 1
Suicidal ideas (Psychiatric disorders) | 1
Fever (General disorders) | 1
Acid reflux (Gastrointestinal disorders) | 1
Ataxia (Nervous system disorders) | 1
Belching (Gastrointestinal disorders) | 1
Hand pain (Musculoskeletal and connective tissue disorders) | 1
Lip picking (Psychiatric disorders) | 1
Paresthesia (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 1
Shoulder injury (Musculoskeletal and connective tissue disorders) | 1
Social withdrawal (Psychiatric disorders) | 1
Stuttering (Nervous system disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT04807517/Prot_SAP_000.pdf